CLINICAL TRIAL: NCT03182192
Title: Visualizing Beta Cells in Patients With Hyperinsulinemic Hypoglycemia After Bariatric Surgery
Brief Title: GLP1R-imaging in Hypoglycemia
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Radboud University Medical Center (Other)
Collaborators: Rijnstate Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: NL51854.091.15
Record Dates: First submitted 2017-05-29; First posted 2017-06-09 (Actual); Last update posted 2023-12-08 (Actual); Status verified 2023-11

CONDITIONS: Hypoglycemia
Keywords: Betal cells; Roux- and Y gastic bypass; exendin; GLP1
MeSH Terms: conditions — Hypoglycemia

STUDY DESIGN:
Intervention Model Description: Comparison of patients with hypoglycemia to control patients
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hypoglycemia (Experimental): Patients with hypoglycemia after gastric bypass
  Interventions: Radiation: 68Ga-NODAGA-exendin-4 PET/CT
- Control (Active Comparator): Patients without hypoglycemia after gastric bypass
  Interventions: Radiation: 68Ga-NODAGA-exendin-4 PET/CT

INTERVENTIONS:
Radiation: 68Ga-NODAGA-exendin-4 PET/CT — 68Ga-NODAGA-exendin-4 PET/CT scan

SUMMARY:
Hyperinsulinemic hypoglycemia (HH) is a rare complication that occurs 1 to 5 years after gastric bypass surgery. The underlying mechanism of this complication is not yet completely understood. Changes in hormone levels, such as GLP1 after RYGB, nesidioblastosis or an increase in the number of beta cells may be one of the underlying causes. However, several study results are conflicting and it is hypothesized that the patient population with HH after RYGB is heterogeneous and several underlying causes may be present. In order to differentiate between hyperfunction with normal beta cell mass and a general or localized increase in beta cell mass we aim to compare quantitative 68Ga-exendin-4 PET imaging of the pancreas between patients with and without HH after RYGB. Thereby, investigators aim to increase the insight in the underlying mechanism of HH after RYGB. If different underlying causes can be diagnosed, treatment for HH can be optimized for patients.

DETAILED DESCRIPTION:
Hyperinsulinaemic hypoglycemia after bariatric surgery. Overweight and obesity are an increasing health problem globally and in the Netherlands, about 15% of the population in the Netherlands is obese. Obesity is associated with increased risk of morbidity, such as cardiovascular disease and type 2 diabetes (T2D). Weight loss is the most important intervention in obese patients, reducing obesity related morbidity and increasing life expectancy. Non-invasive weight loss interventions such as diet, lifestyle or medication only have a moderate effect which is short lived. Weight reducing surgery, i.e. bariatric surgery, is the only intervention that leads to persistent weight loss and is superior above conventional treatment. The most performed and preferred bariatric surgery is Roux-en-Y Gastric Bypass (RYGB), which is a food restrictive and malabsorptive procedure. Besides weight loss, metabolic improvement in T2D patients is an additional result after RYGB.

A frequent late complication of RYGB is the dumping syndrome and a rare late complication is hyperinsulinaemic hypoglycemia (HH). Reported incidences of dumping syndrome range from 20 to 70% of the patients. Dumping is a condition where food enters the small bowel too rapidly and can be divided into early and late dumping. Early dumping is due to rapid gastric emptying and comprises intestinal and vasomotor symptoms within minutes after food ingestion. Late dumping occurs 1 to 3 hours after a meal and the symptoms are partly caused by hypoglycemia.

Reported incidences of HH range from 0.2 to 1% after RYGB and is observed after gastric bypass procedures only. In HH plasma glucose concentrations reach values below 50 mg/dL (2.8 mmol/L) and adrenergic and neuroglucopenic symptoms occur, often occurring after a meal. After a meal or glucose challenge an early large glucose peak followed by an insulin peak is observed in HH patients. Additionally, an increased postprandial GLP1 level compared to RYGB controls without HH was observed. Low plasma glucose levels are also found in asymptomatic patients after RYGB in 30 to 50% of the patients.

The underlying mechanism of HH is not completely understood and several potential causes have been proposed, including, 1) An inappropriate increase of beta cell mass and function, that is persisting despite the increased insulin sensitivity after RYGB, 2) late dumping syndrome, i.e. an inappropriate insulin secretion following rapid food entry into the small intestine, 3) an inappropriate counter-regulatory glucagon response and 4) post-RYGB an increase in the incretin secretion (GLP1 and GIP).

Besides stimulation of the postprandial insulin secretion, GLP1 may induce beta cell hypertrophy or an increase in the number of beta cells by inhibiting apoptosis and increasing replication. Nesidioblastosis (beta cell hypertrophy, islet hyperplasia and increased beta cell mass) is associated with HH after RYGB in some cases, however, nesidioblastosis was not found in these patients and an overexpression of GLP1-receptors in individual islets was not found.

Proposed treatment options for HH after RYGB include diet therapy with a low-carbohydrate diet, drug therapy to inhibit carbohydrate digestion (acarbose) or to inhibit insulin secretion by beta cells (e.g. diaxozide, octreotide, pasireotide) or surgical treatment by a reconstruction of the gastric bypass or by a partial pancreatectomy. The effectiveness of these therapies vary among patients, we expect that the effectiveness of different treatments depends on the underlying cause of HH.

The different possible underlying mechanisms and different types of treatment suggest diverse causes of HH. In order to increase the insight in these causes and to be able to determine the best treatment for each patient in the future, the underlying cause(s) will be examined first in this study. In previous studies that assessed beta cell mass, only only pathological assessment of pancreas specimens was performed, because in vivo assessment was impossible. The control group was determined from patients undergoing a (partial) pancreatectomy for other diseases or post-mortem. However, ideally the control group would consist of patients who have had RYGB as well, without developing HH.

Recently, it became possible to assess beta cell mass in vivo by SPECT and PET imaging. In this study it is examined if this imaging technique can detect an increase in beta cell mass in patients suffering from persisting HH after RYGB. For this purpose we will compare beta cell mass in patients with and without HH after RYGB. Additionally, beta cell function and postprandial incretin responses will be determined in these subjects.

The results of this pilot study may lead to improved diagnostics and treatment options for persisting HH in bariatric patients in future.

Imaging of beta cells in vivo by GLP-1 receptor imaging by PET For specific non-invasive imaging of beta cells, investogators have developed a highly beta cell-specific radiolabeled exendin-based GLP-1 (glucagon-like peptide-1) analog which, after radiolabeling, can non-invasively be detected in the human body. GLP-1 is an incretin hormone that specifically binds to beta cells and is responsible for post-prandial insulin-secretion. Its specificity for beta cells has been shown and a linear correlation of the beta cell mass and the signal obtained with this tracer has been established.

GLP-1R imaging has been shown to be suitable for imaging of insulin producing pancreatic neuroendocrine tumours (IPPNET). Furthermore, the feasibility of visualization of transplanted beta cells with GLP-1R imaging has been shown by imaging of autologous islets transplanted into muscle.

ELIGIBILITY:
Inclusion Criteria:

All individuals:

* Signed informed consent
* > 18

Additional for matched control group:

* RYGB at least 2 years ago
* Normal glucose levels before and after RYGB
* Score <7 on Sigstad's scoring system
* Individual matched to HH group on age

Exclusion Criteria:

All individuals:

* Anti-diabetic medication in the past 6 months
* Treatment with synthetic exendin in the past 6 months
* Liver failure
* Pregnancy
* Breast feeding
* Kidney failure
* Age < 18
* No signed informed consent

Additional for matched control group:

* Any diabetic history
* Previous diagnosed HH
* Sigstad's dumping score >7

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2016-04-01 (Actual); Primary Completion 2024-07-01 (Estimated); Study Completion 2024-07-01 (Estimated)

PRIMARY OUTCOMES:
Uptake of 68Ga-exendin in the pancreas of patients | 1 year
  Calculating uptake by quantitative image analysis

SECONDARY OUTCOMES:
Correlation of tracer uptake with C-peptide and HbA1c | 1 year
  Correlate tracer uptake with C-peptide and HbA1c in patients

CONTACTS AND LOCATIONS:
Locations (2):
- Netherlands (2):
  - Rijnstate hospital, Arnhem, Gelderland
  - Radboudumc, Nijmegen, Gelderland

IPD SHARING:
Plan to Share IPD: No